CLINICAL TRIAL: NCT06826313
Title: An Open-labeled Phase I Clinical Trial Evaluating the Safety, Tolerability, Biodistribution Characteristics, Biological EEffects, and Initial Efficacy of VRT106 for Injection in the Treatment of Locally Advanced/Metastatic Solid Tumors by Intravenous Administration
Brief Title: A Study of Intravenous VRT106 for Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Virotech Pharmaceutical Co., Ltd. (Industry)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRT106-CN01
Record Dates: First submitted 2025-02-10; First posted 2025-02-13 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumors
Keywords: Solid Tumor; Oncolytic Virus; VRT106

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRT106 for injection (Experimental): VRT106 will be administered through IV drip
  Interventions: Biological: VRT106

INTERVENTIONS:
Biological: VRT106 — Intravenous drip administration

SUMMARY:
A Phase I Study of the Safety and Tolerability of VRT106 Administered Intravenously for Treatment of Patients With Locally Advanced or MetastaticSolid Tumors

DETAILED DESCRIPTION:
To evaluate VRT106 for injection in patients with locally advanced/metastatic solid tumours for safety and tolerability, exploring the maximum tolerated dose (MTD)/maximum administered dose (MAD)/optimal bioavailable dose (OBD) and/or the recommended phase II clinical dose (RP2D) to provide a recommended dose for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the clinical study; fully understand and be informed about the study and sign the ICF; and are willing to follow and have the ability to complete all trial procedures.
2. Males and females are aged at 18-75 years (including borderline values) at the time of signing the ICF, male or female.
3. Subjects are histologically or cytologically confirmed to be intolerable or refractory to the standard systemic treatment.
4. Subjects have at least one measurable lesion.
5. ECOG score of 0 to 28 days prior to first dose of IMP.
6. An expected survival time of ≥ 12 weeks.
7. Have sufficient organ function.
8. Female patients of childbearing potential with a negative serum pregnancy test within 7 days prior to first dose of study drug.
9. Subjects of childbearing potential (males and females) agree to use effective birth control with their partner from signing informed consent to at least 90 days after the last dose.

Exclusion Criteria:

1. Subject has received any antitumor therapy within 4 weeks prior to the first dose of IMP.
2. Subject has previously received oncolytic virus or other gene drug therapy.
3. Subject has received treatment with other unlisted clinical investigational drugs/devices within 4 weeks prior to the first dose of IMP.
4. Subject is known to have an allergic reaction to any of the components of IMP.
5. Women who are breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of VRT106 in Patients with advanced malignanttumors | About 2 years
  To evaluate the safety and tolerability of VRT106 in patients with locally advanced/metastatic solid tumours and to explore the maximum tolerated dose (MTD)/multiple ascending dose (MAD)/optimal biologically active dose (OBD) and/or the recommended phase 2 dose (RP2D), which will provide a recommended dose for subsequent clinical trials.

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China